CLINICAL TRIAL: NCT02385162
Title: Biomarker for Glycogen Storage Diseases - AN INTERNATIONAL, MULTICENTER, EPIDEMIOLOGICAL PROTOCOL
Brief Title: Biomarker for Glycogen Storage Diseases (BioGlycogen)
Acronym: BioGlycogen
Status: Withdrawn | Type: Observational
Why Stopped: Transition to BioMetabol
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BGL 06-2018
Record Dates: First submitted 2015-03-02; First posted 2015-03-11 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Fructose Metabolism, Inborn Errors; Glycogen Storage Disease; Glycogen Storage Disease Type I; Glycogen Storage Disease Type II; Glycogen Storage Disease Type III; Glycogen Storage Disease Type IV; Glycogen Storage Disease Type V; Glycogen Storage Disease Type VI; Glycogen Storage Disease Type VII; Glycogen Storage Disease Type VIII
Keywords: Mucolipidoses; Metabolic Diseases; Lysosomal Storage Diseases
MeSH Terms: conditions — Fructose Metabolism, Inborn Errors; Glycogen Storage Disease; Glycogen Storage Disease Type I; Glycogen Storage Disease Type II; Glycogen Storage Disease Type III; Glycogen Storage Disease Type IV; Glycogen Storage Disease Type V; Glycogen Storage Disease Type VI; Glycogen Storage Disease Type VII; Glycogen Storage Disease Type VIII; Mucolipidoses; Metabolic Diseases; Lysosomal Storage Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Für die Entwicklung neuer Biomarker mittels Massenspektrometrie werden 10ml EDTA-Blut und eine Filterkarte mit Trockenblutspots benötigt. Um die korrekte Diagnose für Glykogenosen bei den Patienten zu beweisen, bei denen bis zum Studieneinschluss noch keine genetische Diagnostik vorlag, werden die entsprechenden Sequenzierungen für den Nachweis der Glykogenosen erfolgen. Die Analysen werden von dem Labor Centogene AG pseudonymisiert durchgeführt.
  CENTOGENE AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Patients with a diagnosis of Glycogen storage diseases based upon biochemical and/or genetic criteria or profound suspicion for Glycogen storage disease

SUMMARY:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Glycogen Storage Diseases from plasma. Testing for clinical robustness, specificity and long-term stability of the biomarker.

DETAILED DESCRIPTION:
Glycogen storage diseases (GSDs) are a group of inherited genetic disorders that cause glycogen to be improperly stored in the body. People with glycogen storage diseases have a buildup of abnormal amounts or types of glycogen in their tissues.

The main types of glycogen storage diseases are categorized by number and name. They include:

People with GSD I may have episodes of low blood sugar (hypoglycemia), usually during periods of fasting, due to the ability to store glycogen but inability to properly release it. People with GSD I typically develop an enlarged liver (hepatomegaly) from the storage of glycogen. Elevations in liver function enzymes, blood fat and cholesterol levels, lactic acid, and uric acid also occur. Additional features of GSD I can include decreased bone density, poor growth, kidney disease, liver adenomas, and delayed puberty. Treatment primarily consists of dietary management to maintain normal blood glucose levels and prevent hypoglycemia. GSD I is further divided into subtypes. GSD Type Ia is caused by a deficiency of glucose-6-phosphatase (G6Pase) primarily in the liver, and GSD Type Ib is caused by a deficiency of glucose-6-phosphate translocase. Many of the symptoms are similar, especially early in life. However, some people with Type Ib are more prone to infections given a weaker immune system. GSD I is caused by a non-working change in either the G6PC gene or the SLC37A4 gene, causing the deficiency of the particular enzyme. GSD I follows autosomal recessive inheritance.

Glycogen Storage Disease Type II [also known as Pompe disease, Acid Maltase Deficiency, Glycogenosis Type II, Acid alpha-Glucosidase Deficiency, Lysosomal alpha-Glucosidase Deficiency] Pompe disease is an inherited and often fatal disorder caused by the deficiency of acid alpha-glucosidase (GAA), an enzyme needed to breakdown glycogen (sugar that is stored for energy) in specialized structures in the body, called lysosomes. Patients with Pompe disease have little or no GAA enzyme activity and cannot breakdown glycogen. The excess glycogen accumulates and is stored in the heart, skeletal muscle and other tissues, causing the progressive symptoms of Pompe disease.Glycogen Storage Disease Type III [also known as Cori disease, Forbes disease, Debrancher enzyme deficiency, Limit Dextrinosis]

ELIGIBILITY:
Inclusion Criteria:

* Informed consent will be obtained from the parents before any study related procedures.
* Patients of both genders older than 2 month
* The patient has a diagnosis of glycogen storage disease or a high-grade suspicion for glycogen storage disease

High-grade suspicion present, if one or more inclusion criteria are valid:

* Positive family anamnesis for glycogen storage disease
* Hypoglycemia
* Growth retardation: short stature, skeletal myopathy
* Hepatomegaly, Splenomegaly
* Myopathy with muscle weakness
* cardiomyopathy

Exclusion Criteria:

* No Informed consent from the parents before any study related procedures
* Patients of both genders younger than 2 month
* No diagnosis of glycogen storage disease or no valid criteria for high-grade suspicion of glycogen storage disease

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of glycogen storage disease or profound suspicion for glycogen storage disease
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Glycogen storage disease using the technique of Mass-spectometry 7,5 ml EDTA blood, saliva tube and a dry blood spot filter card | 24 months
  New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

SECONDARY OUTCOMES:
Testing for clinical robustness, specificity and long-term stability of the biomarker | 36 months
  the goal of the study to identify and validate a new biochemical marker from the blood of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (4):
- Centogene AG, Rostock, Germany
- India (2):
  - Amrita Institute of Medical Sciences & Research Centre, Kochi, Kerala
  - Navi Mumbai Institute of Research In Mental And Neurological Handicap (NIRMAN), Mumbai
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: Undecided